CLINICAL TRIAL: NCT03514537
Title: Use of Autologous Stem/Stromal Cellular Stromal Vascular Fraction (cSVF) In Cases Of Frailty and Aging Processes Using Autologous Stem-Stromal Cell Infusion in Patients With Aging Frailty And Wellness
Brief Title: Autologous Stem/Stromal Cellular Stromal Vascular Fraction (cSVF) In Frailty-Aging Processes
Acronym: GARM-W
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID -19 closed facility and testing of subjects
Sponsor: Healeon Medical Inc (Industry)
Collaborators: Micheal Nissenbaum, MD (Unknown); Terry, Glenn C., M.D. (Individual)
Responsible Party: Principal Investigator, Robert W. Alexander, MD, FICS, Principal Investigator, Healeon Medical Inc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GARM-Frailty
Record Dates: First submitted 2018-03-26; First posted 2018-05-02 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-03

CONDITIONS: Frail Elderly Syndrome; Aging; Degenerative Disease
MeSH Terms: interventions — Liberase; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Lipoaspiration (Experimental): Closed microcannula harvesting of small volume of subdermal adipose tissue, including the stromal cellular and stromal tissue using sterile, disposable, microcannula system
  Interventions: Procedure: Microcannula harvest adipose stromal tissues
- Isolation & Concentration of cSVF (Experimental): Isolation and Concentration of cellular stromal vascular fraction (cSVF) using a Healeon Medical CentriCyte 1000 centrifuge, incubator and shaker plate with sterile Liberase enzyme (Roche Medical) per manufacturer protocols
  Interventions: Device: Centricyte 1000; Drug: Liberase
- Delivery cSVF via Intravenous (Experimental): cSVF from Arm 2 is suspended in a 500cc of sterile Normal Saline and deployed through 150 micron in-line filtration and intravenous route over 30-60 minute time frame.
  Interventions: Procedure: Sterile Normal Saline IV Deployment of cSVF; Drug: Saline Solution

INTERVENTIONS:
Procedure: Microcannula harvest adipose stromal tissues — Use of disposable, closed syringe microcannula harvest autologous adipose stroma and stem/stromal cells
  Arms: Lipoaspiration
Device: Centricyte 1000 — Centricyte 1000, closed system digestion of stromal vascular fraction to isolate and concentrate stem/stromal cells associated with microvasculature
  Arms: Isolation & Concentration of cSVF
Procedure: Sterile Normal Saline IV Deployment of cSVF — Sterile Normal Saline Suspension cSVF in 500 cc for Intravenous Delivery including 150 micron in-line filtration
  Arms: Delivery cSVF via Intravenous
Drug: Liberase — Liberase TM for use to enzymatically isolate cellular stromal vascular fraction
  Arms: Isolation & Concentration of cSVF
Drug: Saline Solution — Sterile, Normal Saline 500 for Intravenous use
  Arms: Delivery cSVF via Intravenous

SUMMARY:
With increasing age and health issues associated with aging, many systemic cellular and structural changes are known to occur. The intent of this trial is to determine the safety and efficacy of delivery of autologous cellular stromal vascular fraction (cSVF) to improve the quality of life and functional health.

Isolation and concentration of cSVF will be documented.

To acquire autologous cSVF, a 10+ teaspoon volume of subdermal adipose (fat) tissue and stroma is removed from the trunk or upper thigh area. Using a closed system with enzymatic digestion to isolate and concentrate these cells, is followed with returning these cSVF elements only via 500 cc Normal Saline delivered via peripheral vein (IV).

Documentation of cellular numbers and flow cytometer viability testing is to be correlated with clinical outcomes as reported by patients and standardized Quality of Life (QoL) form tracking

DETAILED DESCRIPTION:
With increasing age and health issues associated with aging, many systemic cellular and structural changes are known to occur. The intent of this trial is to determine the safety and efficacy of delivery of autologous cellular stromal vascular fraction (cSVF) to improve the quality of life and functional health.

Isolation and concentration of cSVF will be documented.

To acquire autologous cSVF, a 10+ teaspoon volume of subdermal adipose (fat) tissue and stroma is removed from the trunk or upper thigh area. Using a closed system with enzymatic digestion to isolate and concentrate these cells, is followed with returning these cSVF elements only via 500 cc Normal Saline delivered via peripheral vein (IV).

Documentation of cellular numbers and flow cytometer viability testing is to be correlated with clinical outcomes as reported by patients and standardized Quality of Life (QoL) form tracking.

Safety of use of certain allogeneic human mesenchymal stem cells (hMSC) has been tested and established along with the effectiveness of use. Autologous stem-stromal cells have been proven safe and effective in many applications and in clinical trials currently underway. These cells are easily obtained and isolated/concentrated in a closed system from patient's adipose derived stromal vascular fraction (cSVF). This is important as such tissues are uniquely the patient's cells, without the need for culture expansion of non-self human tissues, therefore potentially increasing availability to obtain non-allergenic, autologous cells known to be multipotent (can form a variety of specialized cell populations from the body) cell group within the cellular stromal vascular fraction (cSVF) present in essentially all tissues throughout the body (muscle, brain, bone, cartilage, nerve, skin, cardiac muscle, etc.).

This study seeks to determine the safety, efficiency, and in subsequent studies (phase III type) to determine optimal dosages that are needed. Delivery of the cSVF will be returned to the patient's via a standard Normal Saline intravenous infusion (IV).

ELIGIBILITY:
Inclusion Criteria:

* Be >40 and <90 years of age and willing and able to provide written informed consent
* Those aging and frail patients who have noted compromise to activities or work requirements due to increasing age
* Ability to execute a 6 minute walk test distance of >200 meters and <1000 meters
* Loss of energy and exercise tolerance over 6 month period minimum
* Current clinical history of malignancy within 3 years, except for curable skin lesions including basal cell carcinoma, or squamous cell carcinoma
* Must have the ability to provide Informed Consent

Exclusion Criteria:

* Medical conditions which prevent the ability of assessment of walk distance testing criteria
* Have disabling neurodegenerative disorder which would impede interpretation of outcomes
* Have a score of <24 on the Mini Mental State Examination (MMSE)
* History of malignancy within 2 years (excluding curative skin lesion of basal cell carcinoma, melanoma-in-situ, or cervical carcinoma
* Have clinically important abnormal screening laboratory values, including, but not limited to: Hemoglobin <10 g/dL; White blood cell count (WBC) <2500/mL; Platelet count microliters <100000/uL(microliters); Genetic Coagulopathy history
* Uncontrollable hypertension
* Systemic disorders that preclude completion of the testing or out of medical management control in the opinion of the PIs or Primary Care Provider
* Expected lifespan of less that 6 months
* Current drug abuse history < 6 months
* Alcohol abuse within 6 months of enrollment
* Serious or life threatening co-morbidities that in the opinion of investigators, may compromise the safety or compliance with the study guidelines and tracking.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 6 months
  Number of Participants with Treatment Related Adverse & Severe Adverse Events Assessed By CTCAE v4.0

SECONDARY OUTCOMES:
Changes in Weight In Pounds | Baseline and 6 months
  Baseline values at baseline and 6 months;
Activity Level | baseline and 6 months
  Activity level Community Healthy Activities Model Program for Seniors (CHAMPS); Questionnaire; Self Reporting Assessment frequency and duration of various standing, walking, exercise tolerance, and changes in physical activity levels
Mobility | baseline and 6 months
  4 meter gait speed test and short physical performance battery (SPPB); Score of <10 at baseline to predict ability to walk 400 meters
Fatigue | baseline and 6 months
  Multidimensional Fatigue Inventory Questionnaire (MFI); 20 Item self-reporting general fatigue, mental fatigue, reduced motivation, reduced activity levels
Mobility Performance Battery | baseline and 6 months
  Short Mobility Performance Battery (SPPB) Assessment; Evaluates lower extremity function via standing balance (time), 4 meter gait speed and 5 repetition sit to stand (ability)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Nissenbaum, MD, Principal Investigator — Healeon Medical
Locations (1):
- Fanny Island Campus Medical Building, Colchester, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Walston J, Hadley EC, Ferrucci L, Guralnik JM, Newman AB, Studenski SA, Ershler WB, Harris T, Fried LP. Research agenda for frailty in older adults: toward a better understanding of physiology and etiology: summary from the American Geriatrics Society/National Institute on Aging Research Conference on Frailty in Older Adults. J Am Geriatr Soc. 2006 Jun;54(6):991-1001. doi: 10.1111/j.1532-5415.2006.00745.x. PMID 16776798
- [Background] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Background] Song X, Mitnitski A, Rockwood K. Prevalence and 10-year outcomes of frailty in older adults in relation to deficit accumulation. J Am Geriatr Soc. 2010 Apr;58(4):681-7. doi: 10.1111/j.1532-5415.2010.02764.x. Epub 2010 Mar 22. PMID 20345864
- [Background] Lopez-Otin C, Blasco MA, Partridge L, Serrano M, Kroemer G. The hallmarks of aging. Cell. 2013 Jun 6;153(6):1194-217. doi: 10.1016/j.cell.2013.05.039. PMID 23746838
- [Background] Rockwood K, Mitnitski A. Frailty defined by deficit accumulation and geriatric medicine defined by frailty. Clin Geriatr Med. 2011 Feb;27(1):17-26. doi: 10.1016/j.cger.2010.08.008. PMID 21093719
- [Background] Xue QL. The frailty syndrome: definition and natural history. Clin Geriatr Med. 2011 Feb;27(1):1-15. doi: 10.1016/j.cger.2010.08.009. PMID 21093718
- [Background] Tompkins BA, DiFede DL, Khan A, Landin AM, Schulman IH, Pujol MV, Heldman AW, Miki R, Goldschmidt-Clermont PJ, Goldstein BJ, Mushtaq M, Levis-Dusseau S, Byrnes JJ, Lowery M, Natsumeda M, Delgado C, Saltzman R, Vidro-Casiano M, Da Fonseca M, Golpanian S, Premer C, Medina A, Valasaki K, Florea V, Anderson E, El-Khorazaty J, Mendizabal A, Green G, Oliva AA, Hare JM. Allogeneic Mesenchymal Stem Cells Ameliorate Aging Frailty: A Phase II Randomized, Double-Blind, Placebo-Controlled Clinical Trial. J Gerontol A Biol Sci Med Sci. 2017 Oct 12;72(11):1513-1522. doi: 10.1093/gerona/glx137. PMID 28977399
- [Background] Peffers MJ, Collins J, Loughlin J, Proctor C, Clegg PD. A proteomic analysis of chondrogenic, osteogenic and tenogenic constructs from ageing mesenchymal stem cells. Stem Cell Res Ther. 2016 Sep 14;7(1):133. doi: 10.1186/s13287-016-0384-2. PMID 27624072
- [Background] Sethe S, Scutt A, Stolzing A. Aging of mesenchymal stem cells. Ageing Res Rev. 2006 Feb;5(1):91-116. doi: 10.1016/j.arr.2005.10.001. Epub 2005 Nov 28. PMID 16310414
- [Background] Stolzing A, Jones E, McGonagle D, Scutt A. Age-related changes in human bone marrow-derived mesenchymal stem cells: consequences for cell therapies. Mech Ageing Dev. 2008 Mar;129(3):163-73. doi: 10.1016/j.mad.2007.12.002. Epub 2007 Dec 17. PMID 18241911
- [Background] Golpanian S, DiFede DL, Khan A, Schulman IH, Landin AM, Tompkins BA, Heldman AW, Miki R, Goldstein BJ, Mushtaq M, Levis-Dusseau S, Byrnes JJ, Lowery M, Natsumeda M, Delgado C, Saltzman R, Vidro-Casiano M, Pujol MV, Da Fonseca M, Oliva AA Jr, Green G, Premer C, Medina A, Valasaki K, Florea V, Anderson E, El-Khorazaty J, Mendizabal A, Goldschmidt-Clermont PJ, Hare JM. Allogeneic Human Mesenchymal Stem Cell Infusions for Aging Frailty. J Gerontol A Biol Sci Med Sci. 2017 Oct 12;72(11):1505-1512. doi: 10.1093/gerona/glx056. PMID 28444181
- [Background] Hare JM, Traverse JH, Henry TD, Dib N, Strumpf RK, Schulman SP, Gerstenblith G, DeMaria AN, Denktas AE, Gammon RS, Hermiller JB Jr, Reisman MA, Schaer GL, Sherman W. A randomized, double-blind, placebo-controlled, dose-escalation study of intravenous adult human mesenchymal stem cells (prochymal) after acute myocardial infarction. J Am Coll Cardiol. 2009 Dec 8;54(24):2277-86. doi: 10.1016/j.jacc.2009.06.055. PMID 19958962
- [Background] Hare JM, DiFede DL, Rieger AC, Florea V, Landin AM, El-Khorazaty J, Khan A, Mushtaq M, Lowery MH, Byrnes JJ, Hendel RC, Cohen MG, Alfonso CE, Valasaki K, Pujol MV, Golpanian S, Ghersin E, Fishman JE, Pattany P, Gomes SA, Delgado C, Miki R, Abuzeid F, Vidro-Casiano M, Premer C, Medina A, Porras V, Hatzistergos KE, Anderson E, Mendizabal A, Mitrani R, Heldman AW. Randomized Comparison of Allogeneic Versus Autologous Mesenchymal Stem Cells for Nonischemic Dilated Cardiomyopathy: POSEIDON-DCM Trial. J Am Coll Cardiol. 2017 Feb 7;69(5):526-537. doi: 10.1016/j.jacc.2016.11.009. Epub 2016 Nov 14. PMID 27856208
- [Background] Weiss DJ, Casaburi R, Flannery R, LeRoux-Williams M, Tashkin DP. A placebo-controlled, randomized trial of mesenchymal stem cells in COPD. Chest. 2013 Jun;143(6):1590-1598. doi: 10.1378/chest.12-2094. PMID 23172272
- [Background] Karantalis V, Hare JM. Use of mesenchymal stem cells for therapy of cardiac disease. Circ Res. 2015 Apr 10;116(8):1413-30. doi: 10.1161/CIRCRESAHA.116.303614. PMID 25858066
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Golpanian S, DiFede DL, Pujol MV, Lowery MH, Levis-Dusseau S, Goldstein BJ, Schulman IH, Longsomboon B, Wolf A, Khan A, Heldman AW, Goldschmidt-Clermont PJ, Hare JM. Rationale and design of the allogeneiC human mesenchymal stem cells (hMSC) in patients with aging fRAilTy via intravenoUS delivery (CRATUS) study: A phase I/II, randomized, blinded and placebo controlled trial to evaluate the safety and potential efficacy of allogeneic human mesenchymal stem cell infusion in patients with aging frailty. Oncotarget. 2016 Mar 15;7(11):11899-912. doi: 10.18632/oncotarget.7727. PMID 26933813
- [Background] McElhaney JE, Effros RB. Immunosenescence: what does it mean to health outcomes in older adults? Curr Opin Immunol. 2009 Aug;21(4):418-24. doi: 10.1016/j.coi.2009.05.023. Epub 2009 Jun 29. PMID 19570667
- [Background] Kawamoto A, Katayama M, Handa N, Kinoshita M, Takano H, Horii M, Sadamoto K, Yokoyama A, Yamanaka T, Onodera R, Kuroda A, Baba R, Kaneko Y, Tsukie T, Kurimoto Y, Okada Y, Kihara Y, Morioka S, Fukushima M, Asahara T. Intramuscular transplantation of G-CSF-mobilized CD34(+) cells in patients with critical limb ischemia: a phase I/IIa, multicenter, single-blinded, dose-escalation clinical trial. Stem Cells. 2009 Nov;27(11):2857-64. doi: 10.1002/stem.207. PMID 19711453
- [Background] Golpanian S, Schulman IH, Ebert RF, Heldman AW, DiFede DL, Yang PC, Wu JC, Bolli R, Perin EC, Moye L, Simari RD, Wolf A, Hare JM; Cardiovascular Cell Therapy Research Network. Concise Review: Review and Perspective of Cell Dosage and Routes of Administration From Preclinical and Clinical Studies of Stem Cell Therapy for Heart Disease. Stem Cells Transl Med. 2016 Feb;5(2):186-91. doi: 10.5966/sctm.2015-0101. Epub 2015 Dec 18. PMID 26683870
- [Background] Schuleri KH, Feigenbaum GS, Centola M, Weiss ES, Zimmet JM, Turney J, Kellner J, Zviman MM, Hatzistergos KE, Detrick B, Conte JV, McNiece I, Steenbergen C, Lardo AC, Hare JM. Autologous mesenchymal stem cells produce reverse remodelling in chronic ischaemic cardiomyopathy. Eur Heart J. 2009 Nov;30(22):2722-32. doi: 10.1093/eurheartj/ehp265. Epub 2009 Jul 8. PMID 19586959
- [Background] Siddiqi S, Sussman MA. Cell and gene therapy for severe heart failure patients: the time and place for Pim-1 kinase. Expert Rev Cardiovasc Ther. 2013 Aug;11(8):949-57. doi: 10.1586/14779072.2013.814830. PMID 23984924
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Enright PL, McBurnie MA, Bittner V, Tracy RP, McNamara R, Arnold A, Newman AB; Cardiovascular Health Study. The 6-min walk test: a quick measure of functional status in elderly adults. Chest. 2003 Feb;123(2):387-98. doi: 10.1378/chest.123.2.387. PMID 12576356
- [Background] Stewart AL, Mills KM, King AC, Haskell WL, Gillis D, Ritter PL. CHAMPS physical activity questionnaire for older adults: outcomes for interventions. Med Sci Sports Exerc. 2001 Jul;33(7):1126-41. doi: 10.1097/00005768-200107000-00010. PMID 11445760
- [Background] Golpanian S, Wolf A, Hatzistergos KE, Hare JM. Rebuilding the Damaged Heart: Mesenchymal Stem Cells, Cell-Based Therapy, and Engineered Heart Tissue. Physiol Rev. 2016 Jul;96(3):1127-68. doi: 10.1152/physrev.00019.2015. PMID 27335447
- [Background] Rando TA, Wyss-Coray T. Stem cells as vehicles for youthful regeneration of aged tissues. J Gerontol A Biol Sci Med Sci. 2014 Jun;69 Suppl 1(Suppl 1):S39-42. doi: 10.1093/gerona/glu043. PMID 24833585
- [Background] Raggi C, Berardi AC. Mesenchymal stem cells, aging and regenerative medicine. Muscles Ligaments Tendons J. 2012 Oct 16;2(3):239-42. Print 2012 Jul. PMID 23738303
- [Background] Tetta C, Consiglio AL, Bruno S, Tetta E, Gatti E, Dobreva M, Cremonesi F, Camussi G. The role of microvesicles derived from mesenchymal stem cells in tissue regeneration; a dream for tendon repair? Muscles Ligaments Tendons J. 2012 Oct 16;2(3):212-21. Print 2012 Jul. PMID 23738299
- [Background] Alexander, R. Understanding Adipose-derived Stromal Vascular Fraction (AD-SVF) Cell Biology and Use on the Basis of Cellular, Chemical, Structural and Paracrine Components: A Concise Review. J Prolotherapy, 2012 J of Prolo (JOP) 4:e13777
- [Background] Alexander, R., Understanding Mechanical Emulsification (Nanofat) Versus Enzymatic Isolation of Tissue Stromal Vascular Fraction (tSVF) Cells from Adipose Tissue: Potential Uses in Biocellular Regenerative Medicine Understanding J prolo 2016
- [Background] ALEXANDER, ROBERT W., "Biocellular Regenerative Medicine: Adipose-Derived Stem/Stromal Cells & Matrix" . World Biomedical Frontiers, Section of Stem Cells, 2017 July. http://biomedfrontiers.org/stem-cells-2017-7-1.
- [Background] ALEXANDER, ROBERT W., "Use of Microcannula Close Syringe System For Safe And Effective Lipoaspiration and Small Volume Autologous Fat Grafting", Am J Cosm Surg 2013, 30(2): 1-12